CLINICAL TRIAL: NCT03321136
Title: Role of the Serotonin 5-HT2A Receptor in LSD-induced Altered States of Consciousness (LDR-Study)
Acronym: LDR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BASEC-2017-01348
Record Dates: First submitted 2017-09-08; First posted 2017-10-25 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo, LSD-25, LSD-50, LSD-100, LSD-200, LSD-200-Ketanserin (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Placebo
- LSD-25, LSD-50, LSD-100, LSD-200, LSD-200-Ketanserin, Placebo (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Placebo
- LSD-50, LSD-100, LSD-200, LSD-200-Ketanserin, Placebo, LSD-25 (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Placebo
- LSD-100, LSD-200, LSD-200-Ketanserin, Placebo, LSD-25, LSD-50 (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Placebo
- LSD-200, LSD-200-Ketanserin, Placebo, LSD-25, LSD-50, LSD-100 (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Placebo
- LSD-200-Ketanserin, Placebo, LSD-25, LSD-50, LSD-100, LSD-200 (Placebo Comparator): Cross-over within-subjects design with all treatment conditions, separated by a wash-out phase
  Interventions: Drug: LSD; Drug: Placebo

INTERVENTIONS:
Drug: LSD — 0.025 mg LSD per os, single dose
  Other Names: Lysergic Acid Diethylamide
Drug: LSD — 0.05 mg LSD per os, single dose
  Other Names: Lysergic Acid Diethylamide
Drug: LSD — 0.1 mg LSD per os, single dose
  Other Names: Lysergic Acid Diethylamide
Drug: LSD — 0.2 mg LSD per os, single dose
  Other Names: Lysergic Acid Diethylamide
Drug: LSD — 0.2 mg LSD plus 40 mg ketanserin per os, single doses each
  Other Names: Lysergic Acid Diethylamide
Drug: Placebo — Capsules containing mannitol looking identical to the other drugs.

SUMMARY:
Serotonin receptors, especially the 5HT2A receptor, are thought to be involved in the effects of various recreationally used psychedelic substances such as LSD. LSD potently stimulates the 5-HT2A receptor but also 5-HT2B/C, 5-HT1 and dopaminergic receptors. LSD induces acute transient alterations in waking consciousness including visual perceptual alterations, audio-visual synesthesia, derealization and depersonalization. LSD has therefore been used as experimental tool ("psychotomimetic") in modern psychiatric research to study psychotic-like states and model psychosis in healthy subjects [1-5]. However, the dose-effects of 5-HT2A receptor stimulation by LSD has not yet been studied. Additionally, there is still very limited data to what extent the 5HT2A receptor contributes to LSD's effects and its role in the mediation of the full response to LSD at a high dose is unclear. A recent experimental human study showed the 5-HT2A receptor antagonist ketanserin fully blocked the subjective effects of a moderate dose of 100 µg of LSD [6]. But, whether the effects of a high 200 µg oral dose of LSD can be blocked by the selective pharmacological 5-HT2A antagonist ketanserin remains to be tested to confirm the critical role of the 5-HT2A receptor in more pronounced alterations of consciousness and perception. The present study therefore explores the role the 5-HT2A receptor in LSD-induced altered states of consciousness using escalating doses of LSD and the 5-HT2A receptor blocker ketanserin administered before a high dose of LSD.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years.
2. Understanding of the German language.
3. Understanding the procedures and the risks associated with the study.
4. Participants must be willing to adhere to the protocol and sign the consent form.
5. Participants must be willing to refrain from taking illicit psychoactive substances during the study.
6. Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drink after midnight of the evening before the study session, as well as during the study day.
7. Participants must be willing not to drive a traffic vehicle or to operate machines within 48 h after substance administration.
8. Women of childbearing potential must have a negative pregnancy test at the beginning of the study. Pregnancy tests are repeated before each study session.
9. Women of childbearing potential must be willing to use double-barrier birth control
10. Body mass index 18-29 kg/m2.

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder in first-degree relatives
4. Illicit substance use (with the exception of cannabis) more than 10 times or any time within the previous two months.
5. Pregnant or nursing women.
6. Participation in another clinical trial (currently or within the last 30 days)
7. Use of medications that may interfere with the effects of the study medications (any psychiatric medications)
8. Tobacco smoking (>10 cigarettes/day)
9. Consumption of alcoholic drinks (>10/week)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Altered states of consciousness | 18 months
  total 5D-ASC score (5-Dimensional Altered States of Consciousness Rating Scale)

SECONDARY OUTCOMES:
Subjective effects | 18 months
  VAS (Visual analog scales)
Subjective effects | 18 months
  AMRS scales (Adjective mood rating scale)
Psychotomimetic effects | 18 months
  ESI scale (Eppendorf Schizophrenia Inventory)
Mystical-type experiences | 18 months
  MS scales (Mysticism scale)
Mystical-type experiences | 18 months
  SCQ scales (States of consciousness questionnaire)
Autonomic effects | 18 months
  Blood pressure
Autonomic effects | 18 months
  Heart Rate
Autonomic effects | 18 months
  Body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No